CLINICAL TRIAL: NCT00242632
Title: Cognitive Effects of Memantine in Postmenopausal Women at Risk of Dementia: a Pilot Study
Brief Title: Treatment With Namenda in Women at Risk for Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Natalie Rasgon, Principal Investigator, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 95239
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ApoE Non-Carriers (Experimental): Subjects in this group did not carry the apolipoprotein E-epsilon 4 (apoE-e4) allele. During week 1 of the study, subjects were administered 5 mg of namenda once daily. During week 2 of the study, subjects were administered 5 mg of namenda in the morning and 5 mg in the evening (10 mg/day). During week 3 of the study, subjects were administered 10 mg in the morning and 5 mg in the evening (15 mg/day). During week 4 of the study, subjects were administered 10 mg in the morning and 10 mg in the evening (20 mg/day).
  Interventions: Drug: Namenda
- ApoE Carriers (Experimental): Subjects in this group carried the apolipoprotein E-epsilon 4 (apoE-e4) allele. During week 1 of the study, subjects were administered 5 mg of namenda once daily. During week 2 of the study, subjects were administered 5 mg of namenda in the morning and 5 mg in the evening (10 mg/day). During week 3 of the study, subjects were administered 10 mg in the morning and 5 mg in the evening (15 mg/day). During week 4 of the study, subjects were administered 10 mg in the morning and 10 mg in the evening (20 mg/day).
  Interventions: Drug: Namenda

INTERVENTIONS:
Drug: Namenda — Namenda has already been shown to offer cognitive benefits to patients suffering from Alzheimer's disease, but it's potential for treating those at risk for cognitive decline without Alzheimer's disease or other dementia has yet to be evaluated. It is possible that memantine may offer neurocognitive benefits to this population, as well. Participants are asked to take medication for six months, complete neuropsychological testing, and one blood draw.
  Other Names: Memantine

SUMMARY:
This research aims to explore the effectiveness of memantine (Namenda) in treating post-menopausal women between the ages of 50 and 65, who are at risk for cognitive decline. Memantine has already been shown to offer cognitive benefits to patients suffering from Alzheimer's disease, but it's potential for treating those at risk for cognitive decline without Alzheimer's disease or other dementia has yet to be evaluated. It is possible that memantine may offer neurocognitive benefits to this population, as well. Participants are asked to take medication for six months, complete neuropsychological testing, and one blood draw.

DETAILED DESCRIPTION:
Memantine is a well-tolerated moderate-affinity, uncompetitive, voltage-dependent NMDA receptor antagonist that is shown to improve cognition and behavior in mild to moderate and moderate to severe Alzheimer's disease (AD). More recent, albeit limited, evidence also shows benefits of memantine treatment in a host of other disorders such as vascular dementia, pervasive developmental disorders, depression and frontal temporal dementia case studies. However, no studies to date have sought to determine if memantine has potential as a primary prevention for AD.

Incidence rates of AD are expected to more than double from 1995 to the year 2050 as baby boomers age and it is predicted that this substantial increase will create a devastating global burden. At present, there are no treatments that prevent or 'cure' AD; however, treatments that delay the onset of dementia could provide significant reductions in incident rates. Epidemiological studies estimate that an increase in cognitive reserve of only 5% would substantially reduce the incidence rate of AD by one-third; therefore, interventions that precede the manifestation of AD would be most beneficial.

Over the past several years, research on dementia focused on determining the factors that were involved in the progression from mild cognitive impairment to dementia. Clearly, when interventions can be introduced before any cognitive decline is evident the better the chance of reducing incidence dementia. Few studies have investigated risk factors for AD other than genetic vulnerability and primary prevention studies are essentially non-existent. Known and putative risk factors for AD include being a carrier of an apolipoprotein E-epsilon 4 (apoE-ɛ4) allele, particularly for late-onset AD, family history of AD, history of depression, hypothyroidism, and diabetes. This study was a prospective open-label, 6-month pilot medication trial to determine potential salutary effects of memantine on cognition in women at risk of AD. The study design included built-in control for the genetic risk factor for AD (apoE-ɛ4 status). In addition, this study sought to determine whether memantine administration could provide any cognitive benefits to a population of normal postmenopausal women with at least one other putative risk factor for AD.

ELIGIBILITY:
Inclusion Criteria::

* Women between the ages of 50-65
* Willing to sign Human Subjects Protection Consent Form
* Personal or family history of mood disorder
* Hypothyroidism
* Diabetes
* Family history of Alzheimer's disease Exclusion Criteria:- Possible or probable Alzheimer's disease or dementia
* History of cerebrovascular disease
* History of myocardial infarction within the previous year
* History of unstable heart disease
* Uncontrolled hypertension
* Less than 8 years of education
* English as a 2nd language
* Uncorrected vision or hearing deficits

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Natalie Rasgon, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- apoE-e4-: Subjects without the apoE-e4 allele
- apoE-e4+: Subjects with the apoE-e4 allele
Period: Overall Study
Arm/Group | apoE-e4- | apoE-e4+
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | apoE-e4- | apoE-e4+ | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.73 (0) | 59.09 (0) | 58.41 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in California Verbal Learning Test - Second Edition Proactive Interference Test Between Time 1 and Time 2
Description: This tests verbal memory (word list). A list of words is presented and subjects are asked to recall as many as they can. Then a list of interference words is presented. Finally a recognition list of 44 words is presented where subjects are asked to distinguish between target words and distractors. The mean difference in the percentage of target words recalled between time 1 and time 2 is calculated below.
Time Frame: 6 months
Population: All participants were grouped together for this Outcome Measure. As per the protocol, the analyses of neuropsychological variables were to be done separately for the ApoE-ɛ4 carriers and non-carriers, only if the ApoE-ε4 status was a significant predictor of change in neuropsychological performance.
Measure: Mean (Standard Deviation); unit: percentage of target words recalled
Groups:
- T1-T2: This arm includes all 22 subjects from Time 1 to Time 2, a 6-month period.
Arm/Group | T1-T2
Number analyzed (Participants) | 22
percentage of target words recalled | 20.41 (5.63)

2. Secondary Outcome: Change in Delis-Kaplan Executive Function System (DKEFS) Verbal Fluency Category Switching Between Time 1 and Time 2
Description: The Delis-Kaplan Executive Function System (DKEFS) Verbal Fluency Category Switching test measures letter fluency, category fluency, and category switching. The score is the total number of correct words generated during each of the 60-second trials within the three conditions of the test. The mean difference in the total number of correct words generated between time 1 and time 2 is calculated below.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: correct words
Arm/Group | T1-T2
Number analyzed (Participants) | 22
correct words | 1.11 (0.23)

ADVERSE EVENTS:
Time Frame: The time period was 6 months.
Groups:
- ApoE-e4+: This includes the 11 subjects who were carriers of the ApoE-e4 allele.
- ApoE-e4-: This includes the 11 subjects who were non-carriers of the ApoE-e4 allele.
Arm/Group | ApoE-e4+ | ApoE-e4-
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No